CLINICAL TRIAL: NCT01185626
Title: ROGYcare: The Impact of a Cancer Survivorship Care Plan on Patient Reported Outcomes and Health Care Providers. A Pragmatic Cluster Randomized Controlled Trial
Brief Title: ROGYcare: The Impact of a Cancer Survivorship Care Plan on Patient Reported Outcomes and Health Care Providers
Acronym: ROGYcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lonneke van de Poll-Franse (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other); Dutch Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Lonneke van de Poll-Franse, Dr. Prof., Tilburg University
Organization: Tilburg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UVT 2010-4743
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer; Endometrium Cancer
Keywords: patients
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): The gynaecological oncologist (GO) provides care as usual. Currently, hospitals provide follow-up following the Dutch guidelines, meaning that they see their patients on given time points based on the number of years after diagnosis. Most hospitals give their patients leaflets regarding the diagnosis and treatment they receive, however none of them provide personalized information. All information is given during the initial treatment phase, but none of the GOs give additional information during follow-up. None of the GOs is actively screening on psychosocial needs. As this might change in time, we will ask the providers and patients about the type of information they provide, respectively, receive.
- SCP care (Experimental): After initial treatment, the GO provides the patient with a paper SCP and takes time to discuss all items in the SCP. Each time during follow-up meetings between patient and GO, the patient will receive an updated SCP if applicable. The paper SCP is extracted from the online registration system 'ROGY' (Registrationsystem Oncological GYnaecology) and combines personal patient and disease data with tailored information that is related to the specific situation of this patient. Recurrences, toxicities or additionally involved specialists will be registered in ROGY and automatically updated in the personal SCP.
  Interventions: Other: SCP care

INTERVENTIONS:
Other: SCP care
  Arms: SCP care

SUMMARY:
Earlier diagnoses and improved treatments have contributed to the growing cohort of cancer survivors. Nevertheless, these patients remain at risk for adverse long-term or late physical or psychosocial effects of cancer and its treatment. There is increasing recognition to improve information disclosure and cancer survivorship care. The American Institute of Medicine (IOM) and Health Council of the Netherlands both recommend that cancer survivors receive a summary of their course of treatment as a formal document, that also includes recommendations for subsequent cancer surveillance, management of late effects, and strategies for health promotion, the Survivorship Care Plan (SCP). However, no evidence exists concerning the positive and negative effects of the implementation of the SCP in daily clinical practice. The purpose of this study is to assess the impact of SCP care in routine clinical practice on cancer survivors' satisfaction with information disclosure and care, quality of life, illness perception, and health care use.

ELIGIBILITY:
Inclusion Criteria:

* Women who are newly diagnosed with endometrial or ovarian cancer in one of the 12 participating hospitals.
* The patients have to be able to complete a Dutch questionnaire.

Exclusion Criteria:

* Patients who are not able to read or write Dutch will be excluded, as they are not able to complete a Dutch questionnaire.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Patients' score on the EORTC-INFO26 module15 questionnaire, measuring ´Satisfaction with information provision´, right after initial treatment | Right after initial treatment (t0)
  Evaluating satisfaction with information on different areas of the disease, diagnosis, treatment and care. It contains the following scales: (a) Information about the disease; (b) Information about medical tests; (c) Information about treatment; (d) Information on other services, and single items: (a) Written information; (b) Information on CDs or tape/video; (c) Satisfaction with the amount of information; (d) Desire for more information; (e) Desire for less information; (f) Helpfulness of information.
Patients' score on the EORTC QLQ-C3017 questionnaire, measuring ´Health related quality of life (HRQL)´, right after initial treatment | Right after initial treatment (t0)
  Measuring cancer specific HRQL, including scales assessing physical, role, cognitive and emotional functioning, fatigue and sleep problems, and overall health and quality of life.This core instrument is supplemented by a condition-specific questionnaire module (for ovarian cancer: EORTC-OV module18, for endometrial cancer: EORTC-EN module).
Patients' score on the EORTC IN-PATSAT3216 questionnaire, measuring ´Satisfaction with care´, right after initial treatment | Right after initial treatment (t0)
  Assessing patients' perception of quality of medical care, nursing care and care organization and hospital services . It contains 11 multi-item and 3 single-item scales, including doctors' and nurses' skills, information provision, and availability.
Patients' score on the Brief Illness Perception Questionnaire (B-IPQ)21, measuring ´Illness perception´, right after initial treatment | Right after initial treatment (t0)
  The scale has 9 items, measuring (a) cognitive representations (consequences, timeline, personal control, treatment control, identity); (b) emotional representations (concern, emotion); (c) illness comprehensibility; and (d) an open-ended response item on the 3 most important causal factors of illness.
Patients' score on the EORTC-INFO26 module15 questionnaire, measuring ´Satisfaction with information provision´, 6 months after initial treatment | 6 months after initial treatment (t1)
  Evaluating satisfaction with information on different areas of the disease, diagnosis, treatment and care. It contains the following scales: (a) Information about the disease; (b) Information about medical tests; (c) Information about treatment; (d) Information on other services, and single items: (a) Written information; (b) Information on CDs or tape/video; (c) Satisfaction with the amount of information; (d) Desire for more information; (e) Desire for less information; (f) Helpfulness of information.
Patients' score on the EORTC QLQ-C3017 questionnaire, measuring ´Health related quality of life (HRQL)´, 6 months after initial treatment | 6 months after initial treatment (t1)
  Measuring cancer specific HRQL, including scales assessing physical, role, cognitive and emotional functioning, fatigue and sleep problems, and overall health and quality of life.This core instrument is supplemented by a condition-specific questionnaire module (for ovarian cancer: EORTC-OV module18, for endometrial cancer: EORTC-EN module).
Patients' score on the EORTC IN-PATSAT3216 questionnaire, measuring ´Satisfaction with care´, 6 months after initial treatment | 6 months after initial treatment (t1)
  Assessing patients' perception of quality of medical care, nursing care and care organization and hospital services . It contains 11 multi-item and 3 single-item scales, including doctors' and nurses' skills, information provision, and availability.
Patients' score on the Brief Illness Perception Questionnaire (B-IPQ)21, measuring ´Illness perception´, 6 months after initial treatment | 6 months after initial treatment (t1)
  The scale has 9 items, measuring (a) cognitive representations (consequences, timeline, personal control, treatment control, identity); (b) emotional representations (concern, emotion); (c) illness comprehensibility; and (d) an open-ended response item on the 3 most important causal factors of illness.
Patients' score on the EORTC-INFO26 module15 questionnaire, measuring ´Satisfaction with information provision´, 12 months after initial treatment | 12 months after initial treatment (t2)
  Evaluating satisfaction with information on different areas of the disease, diagnosis, treatment and care. It contains the following scales: (a) Information about the disease; (b) Information about medical tests; (c) Information about treatment; (d) Information on other services, and single items: (a) Written information; (b) Information on CDs or tape/video; (c) Satisfaction with the amount of information; (d) Desire for more information; (e) Desire for less information; (f) Helpfulness of information.
Patients' score on the EORTC QLQ-C3017 questionnaire, measuring ´Health related quality of life (HRQL)´, 12 months after initial treatment | 12 months after initial treatment (t2)
  Measuring cancer specific HRQL, including scales assessing physical, role, cognitive and emotional functioning, fatigue and sleep problems, and overall health and quality of life.This core instrument is supplemented by a condition-specific questionnaire module (for ovarian cancer: EORTC-OV module18, for endometrial cancer: EORTC-EN module).
Patients' score on the EORTC IN-PATSAT3216 questionnaire, measuring ´Satisfaction with care´, 12 months after initial treatment | 12 months after initial treatment (t2)
  Assessing patients' perception of quality of medical care, nursing care and care organization and hospital services . It contains 11 multi-item and 3 single-item scales, including doctors' and nurses' skills, information provision, and availability.
Patients' score on the Brief Illness Perception Questionnaire (B-IPQ)21, measuring ´Illness perception´, 12 months after initial treatment | 12 months after initial treatment (t2)
  The scale has 9 items, measuring (a) cognitive representations (consequences, timeline, personal control, treatment control, identity); (b) emotional representations (concern, emotion); (c) illness comprehensibility; and (d) an open-ended response item on the 3 most important causal factors of illness.
Patients' score on the EORTC-INFO26 module15 questionnaire, measuring ´Satisfaction with information provision´, 18 months after initial treatment | 18 months after initial treatment (t3)
  Evaluating satisfaction with information on different areas of the disease, diagnosis, treatment and care. It contains the following scales: (a) Information about the disease; (b) Information about medical tests; (c) Information about treatment; (d) Information on other services, and single items: (a) Written information; (b) Information on CDs or tape/video; (c) Satisfaction with the amount of information; (d) Desire for more information; (e) Desire for less information; (f) Helpfulness of information.
Patients' score on the EORTC QLQ-C3017 questionnaire, measuring ´Health related quality of life (HRQL)´, 18 months after initial treatment | 18 months after initial treatment (t3)
  Measuring cancer specific HRQL, including scales assessing physical, role, cognitive and emotional functioning, fatigue and sleep problems, and overall health and quality of life.This core instrument is supplemented by a condition-specific questionnaire module (for ovarian cancer: EORTC-OV module18, for endometrial cancer: EORTC-EN module).
Patients' score on the EORTC IN-PATSAT3216 questionnaire, measuring ´Satisfaction with care´, 18 months after initial treatment | 18 months after initial treatment (t3)
  Assessing patients' perception of quality of medical care, nursing care and care organization and hospital services . It contains 11 multi-item and 3 single-item scales, including doctors' and nurses' skills, information provision, and availability.
Patients' score on the Brief Illness Perception Questionnaire (B-IPQ)21, measuring ´Illness perception´, 18 months after initial treatment | 18 months after initial treatment (t3)
  The scale has 9 items, measuring (a) cognitive representations (consequences, timeline, personal control, treatment control, identity); (b) emotional representations (concern, emotion); (c) illness comprehensibility; and (d) an open-ended response item on the 3 most important causal factors of illness.
Patients' score on the EORTC-INFO26 module15 questionnaire, measuring ´Satisfaction with information provision´, 24 months after initial treatment | 24 months after initial treatment (t4)
  Evaluating satisfaction with information on different areas of the disease, diagnosis, treatment and care. It contains the following scales: (a) Information about the disease; (b) Information about medical tests; (c) Information about treatment; (d) Information on other services, and single items: (a) Written information; (b) Information on CDs or tape/video; (c) Satisfaction with the amount of information; (d) Desire for more information; (e) Desire for less information; (f) Helpfulness of information.
Patients' score on the EORTC QLQ-C3017 questionnaire, measuring ´Health related quality of life (HRQL)´, 24 months after initial treatment | 24 months after initial treatment (t4)
  Measuring cancer specific HRQL, including scales assessing physical, role, cognitive and emotional functioning, fatigue and sleep problems, and overall health and quality of life.This core instrument is supplemented by a condition-specific questionnaire module (for ovarian cancer: EORTC-OV module18, for endometrial cancer: EORTC-EN module).
Patients' score on the EORTC IN-PATSAT3216 questionnaire, measuring ´Satisfaction with care´, 24 months after initial treatment | 24 months after initial treatment (t4)
  Assessing patients' perception of quality of medical care, nursing care and care organization and hospital services . It contains 11 multi-item and 3 single-item scales, including doctors' and nurses' skills, information provision, and availability.
Patients' score on the Brief Illness Perception Questionnaire (B-IPQ)21, measuring ´Illness perception´, 24 months after initial treatment | 24 months after initial treatment (t4)
  The scale has 9 items, measuring (a) cognitive representations (consequences, timeline, personal control, treatment control, identity); (b) emotional representations (concern, emotion); (c) illness comprehensibility; and (d) an open-ended response item on the 3 most important causal factors of illness.

SECONDARY OUTCOMES:
Patients' frequency and reason (cancer-related or not) for contact with their general practitioner or medical specialist in the past 12 months, measuring 'Patients' health care use', right after initial treatment | Right after initial treatment (t0)
  Patients will also be asked whether they have been referred to other health care services.
Health care providers' score on a questionnaire assessing their evaluation of the (implementation of the) SCP | At the start of the study (t0)
  The questionnaire will contain questions regarding how much time the health care providers in general expect to spend on SCP care, and what problems they expect to encounter in daily practice.
Health care providers' score on a questionnaire assessing their evaluation of the (implementation of the) SCP | At the end of the study (t5)
  The questionnaire will contain questions regarding how much time the health care providers spent on SCP care, and what problems they encountered in daily practice.
Patients' frequency and reason (cancer-related or not) for contact with their general practitioner or medical specialist in the past 12 months, measuring 'Patients' health care use', 6 months after initial treatment | 6 months after initial treatment (t1)
  Patients will also be asked whether they have been referred to other health care services.
Patients' frequency and reason (cancer-related or not) for contact with their general practitioner or medical specialist in the past 12 months, measuring 'Patients' health care use', 12 months after initial treatment | 12 months after initial treatment (t2)
  Patients will also be asked whether they have been referred to other health care services.
Patients' frequency and reason (cancer-related or not) for contact with their general practitioner or medical specialist in the past 12 months, measuring 'Patients' health care use', 18 months after initial treatment | 18 months after initial treatment (t3)
  Patients will also be asked whether they have been referred to other health care services.
Patients' frequency and reason (cancer-related or not) for contact with their general practitioner or medical specialist in the past 12 months, measuring 'Patients' health care use', 24 months after initial treatment | 24 months after initial treatment (t4)
  Patients will also be asked whether they have been referred to other health care services.

CONTACTS AND LOCATIONS:
Overall Officials: Lonneke V van de Poll-Franse, Dr. Prof., Principal Investigator — Tilburg University, The Netherlands; Nicole PM Ezendam, Dr., Principal Investigator — The Netherlands Comprehensive Cancer Organisation
Locations (12):
- Netherlands (12):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Amphia Ziekenhuis, Breda
  - Catharina-Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - St. Anna Ziekenhuis, Geldrop
  - Elkerliek Ziekenhuis, Helmond
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Orbis Medisch Centrum, Sittard
  - St. Elisabeth Hospital, Tilburg
  - TweeSteden Ziekenhuis, Tilburg
  - VieCuri Medisch Centrum, Venlo
  - St. Jans Gasthuis, Weert

REFERENCES:
- [Background] van de Poll-Franse LV, Nicolaije KA, Vos MC, Pijnenborg JM, Boll D, Husson O, Ezendam NP, Boss EA, Hermans RH, Engelhart KC, Haartsen JE, Pijlman BM, Feijen HW, Mertens HJ, Nolting WE, van Beek JJ, Roukema JA, Kruitwagen RF. The impact of a cancer Survivorship Care Plan on gynecological cancer patient and health care provider reported outcomes (ROGY Care): study protocol for a pragmatic cluster randomized controlled trial. Trials. 2011 Dec 5;12:256. doi: 10.1186/1745-6215-12-256. PMID 22141750
- [Result] Nicolaije KA, Ezendam NP, Vos MC, Pijnenborg JM, Boll D, Boss EA, Hermans RH, Engelhart KC, Haartsen JE, Pijlman BM, van Loon-Baelemans IE, Mertens HJ, Nolting WE, van Beek JJ, Roukema JA, Zijlstra WP, Kruitwagen RF, van de Poll-Franse LV. Impact of an Automatically Generated Cancer Survivorship Care Plan on Patient-Reported Outcomes in Routine Clinical Practice: Longitudinal Outcomes of a Pragmatic, Cluster Randomized Trial. J Clin Oncol. 2015 Nov 1;33(31):3550-9. doi: 10.1200/JCO.2014.60.3399. Epub 2015 Aug 24. PMID 26304900
- [Result] Ezendam NP, Nicolaije KA, Kruitwagen RF, Pijnenborg JM, Vos MC, Boll D, van Bommel M, van de Poll-Franse LV. Survivorship Care Plans to inform the primary care physician: results from the ROGY care pragmatic cluster randomized controlled trial. J Cancer Surviv. 2014 Dec;8(4):595-602. doi: 10.1007/s11764-014-0368-0. Epub 2014 May 28. PMID 24866923
- [Result] Nicolaije KA, Ezendam NP, Vos MC, Pijnenborg JM, van de Poll-Franse LV, Kruitwagen RF. Oncology providers' evaluation of the use of an automatically generated cancer survivorship care plan: longitudinal results from the ROGY Care trial. J Cancer Surviv. 2014 Jun;8(2):248-59. doi: 10.1007/s11764-013-0327-1. Epub 2013 Dec 20. PMID 24357226
- [Result] Nicolaije KA, Ezendam NP, Pijnenborg JM, Boll D, Vos MC, Kruitwagen RF, van de Poll-Franse LV. Paper-Based Survivorship Care Plans May be Less Helpful for Cancer Patients Who Search for Disease-Related Information on the Internet: Results of the Registrationsystem Oncological Gynecology (ROGY) Care Randomized Trial. J Med Internet Res. 2016 Jul 8;18(7):e162. doi: 10.2196/jmir.4914. PMID 27392550
- [Result] de Rooij BH, Ezendam NP, Nicolaije KA, Vos MC, Pijnenborg JM, Boll D, Kruitwagen RF, van de Poll-Franse LV. Factors influencing implementation of a survivorship care plan-a quantitative process evaluation of the ROGY Care trial. J Cancer Surviv. 2017 Feb;11(1):64-73. doi: 10.1007/s11764-016-0562-3. Epub 2016 Aug 1. PMID 27480883
- [Result] van Broekhoven MECL, de Rooij BH, Pijnenborg JMA, Vos MC, Boll D, Kruitwagen RFPM, van de Poll-Franse LV, Ezendam NPM. Illness perceptions and changes in lifestyle following a gynecological cancer diagnosis: A longitudinal analysis. Gynecol Oncol. 2017 May;145(2):310-318. doi: 10.1016/j.ygyno.2017.02.037. Epub 2017 Mar 6. PMID 28279480
- [Result] de Rooij BH, Ezendam NPM, Nicolaije KAH, Caroline Vos M, Pijnenborg JMA, Boll D, Boss EA, Hermans RHM, Engelhart KCM, Haartsen JE, Pijlman BM, van Loon-Baelemans IEAM, Mertens HJMM, Nolting WE, van Beek JJ, Roukema JA, Kruitwagen RFPM, van de Poll-Franse LV. Effects of Survivorship Care Plans on patient reported outcomes in ovarian cancer during 2-year follow-up - The ROGY care trial. Gynecol Oncol. 2017 May;145(2):319-328. doi: 10.1016/j.ygyno.2017.02.041. Epub 2017 Mar 7. PMID 28283195
- [Derived] Driessen KAJ, de Rooij BH, Vos MC, Boll D, Pijnenborg JMA, Hoedjes M, Beijer S, Ezendam NPM. Cancer-related psychosocial factors and self-reported changes in lifestyle among gynecological cancer survivors: cross-sectional analysis of PROFILES registry data. Support Care Cancer. 2022 Feb;30(2):1199-1207. doi: 10.1007/s00520-021-06433-0. Epub 2021 Aug 28. PMID 34453569
- [Derived] de Rooij BH, Ezendam NPM, Nicolaije KAH, Lodder P, Vos MC, Pijnenborg JMA, Boll D, Kruitwagen RFPM, van de Poll-Franse LV. Survivorship care plans have a negative impact on long-term quality of life and anxiety through more threatening illness perceptions in gynecological cancer patients: the ROGY care trial. Qual Life Res. 2018 Jun;27(6):1533-1544. doi: 10.1007/s11136-018-1825-4. Epub 2018 Mar 6. PMID 29511906